CLINICAL TRIAL: NCT00086892
Title: A Phase II Evaluation of Cetuximab (C225, NSC #714692) in Combination With Carboplatin (NSC #241240) in the Treatment of Recurrent Platinum-Sensitive Ovarian or Primary Peritoneal Cancer
Brief Title: Cetuximab and Carboplatin in Treating Patients With Recurrent Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Masking: None | Purpose: Treatment
Other Study IDs: GOG-0146P; BMS-CA225-019; CDR0000371712
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Cetuximab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: cetuximab
Drug: carboplatin

SUMMARY:
RATIONALE: Monoclonal antibodies such as cetuximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy such as carboplatin work in different ways to stop tumor cells from dividing so they stop growing or die. Combining cetuximab with carboplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with carboplatin works in treating patients with recurrent ovarian epithelial cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of cetuximab and carboplatin in patients with recurrent platinum-sensitive ovarian epithelial or primary peritoneal cancer.
* Determine the nature and degree of toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 1 hour (over 2 hours on day 1 of course 1 only) on days 1, 8 , and 15. Patients also receive carboplatin IV after cetuximab administration on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 20-65 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial or primary peritoneal cancer

  * Recurrent disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques, including palpation, plain x-ray, CT scan, or MRI OR ≥ 10 mm by spiral CT scan
  * Target lesion not within previously irradiated field
* Received 1 prior platinum-based chemotherapy regimen for primary disease containing carboplatin, cisplatin, or other organoplatinum compound

  * Initial treatment may have included high-dose, consolidation, or extended therapy administered after surgical or non-surgical assessment
  * Patients who had not received prior paclitaxel therapy may have received a second regimen that included paclitaxel
* Platinum-sensitive disease

  * Treatment-free interval without clinical evidence of progressive disease for more than 6 months after response to a prior platinum-based regimen
  * If there is another concurrently active GOG-0146 series protocol (non-platinum-based therapy), must have had a treatment-free interval of more than 12 months unless ineligible for the other protocol* NOTE: *Applies whether or not both protocols are available at the same participating center
* Must have available tissue block or unstained sections from primary tumor, interval debulking, or secondary debulking
* Not eligible for a higher priority GOG protocol (i.e., any active phase III GOG protocol for the same patient population)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No uncontrolled hypertension
* No unstable angina
* No congestive heart failure
* No uncontrolled arrhythmias within the past 6 months
* No other significant cardiac disease

Neurologic

* No uncontrolled seizure disorder
* No active neurological disease
* No neuropathy > grade 1

Other

* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No active infection requiring antibiotics
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior anti-epidermal growth factor receptor (EGFR) antibody therapy
* No prior chimerized or murine monoclonal antibody therapy
* At least 3 weeks since prior biologic or immunologic therapy for the malignancy

Chemotherapy

* See Disease Characteristics
* Recovered from prior chemotherapy
* No prior cytotoxic chemotherapy for recurrent disease, including retreatment with initial chemotherapy regimens

Endocrine therapy

* At least 1 week since prior hormonal therapy for the malignancy
* Concurrent hormone replacement therapy allowed

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy
* No prior radiotherapy to > 25% of bone marrow-bearing areas

Surgery

* More than 30 days since prior major surgery and recovered

  * Diagnostic biopsy not considered major surgery

Other

* At least 3 weeks since other prior therapy for the malignancy
* No prior tyrosine kinase inhibitors that target the EGFR pathway
* No prior cancer treatment that would preclude study treatment
* No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angeles A. Secord, MD, Study Chair — Duke Cancer Institute; Deborah K. Armstrong, MD — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Nita Maihle, PhD — Yale University
Locations (76):
- United States (72):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Women's Cancer Center - Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Hinsdale, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Tufts - New England Medical Center, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Cancer Institute of New Jersey at the Cooper University Hospital - Voorhees, Camden, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase-Temple Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Southeast Gynecologic Oncology Associates, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Fletcher Allen Health Care - Medical Center Hospital of Vermont Campus, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Australia New Zealand Gynaecological Oncology Trials Group, Camperdown, New South Wales, Australia
- Tom Baker Cancer Centre - Calgary, Calgary, Alberta, Canada
- Kagoshima City Hospital, Kagoshima, Japan
- Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Result] Secord AA, Blessing JA, Armstrong DK, Rodgers WH, Miner Z, Barnes MN, Lewandowski G, Mannel RS; Gynecologic Oncology Group. Phase II trial of cetuximab and carboplatin in relapsed platinum-sensitive ovarian cancer and evaluation of epidermal growth factor receptor expression: a Gynecologic Oncology Group study. Gynecol Oncol. 2008 Mar;108(3):493-9. doi: 10.1016/j.ygyno.2007.11.029. Epub 2008 Jan 14. PMID 18191993